CLINICAL TRIAL: NCT04827160
Title: Predictive Value of D-dimers Trends and Levels for Thrombosis in Patients With COVID-19
Brief Title: Prediction of Thrombosis Using D-dimer Trends in COVID-19
Acronym: TRENDS
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Stéphane Zuily, Professor, Central Hospital, Nancy, France
Other Study IDs: 2020308
Record Dates: First submitted 2021-03-30; First posted 2021-04-01 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- COVID-19: Patients with COVID-19

SUMMARY:
A high incidence of venous thromboembolic events (VTE) has been demonstrated in COVID-19. This incidence correlates with disease severity. Activation of coagulation secondary to sepsis combined with classical thrombotic risk factors may contribute to this prothrombotic state. Since the beginning of March 2020, the issue of venous thrombosis during SARS-CoV-2 infection has rapidly emerged as a major medical challenge since a significant rate of patients were thrombosing, some of them in spite of a well conducted preventive anticoagulation. Although D-dimers have been shown to be useful in identifying patients at risk of severe COVID-19 and even mortality, they cannot be used for diagnostic exclusion of pulmonary embolism. Indeed, since D-dimer levels rise non-specifically during infectious states, the exclusion threshold of 500 ng/ml cannot be used.

It would therefore be useful to study the predictive value of D-dimers for thrombosis in COVID-19 patients.

DETAILED DESCRIPTION:
Primary outcome : Characterize different D-dimer trends in COVID-19 patients.

Secondary outcomes :

* Identify the predictive value of different D-dimers trends for thrombosis / all-cause mortality / orotracheal intubation during hospitalization
* Identify the predictive value of D-dimers at admission for thrombosis / all-cause mortality / orotracheal intubation during hospitalization
* Identify the predictive value of 1st D-dimer/fibrinogen ratio for thrombosis / all-cause mortality / orotracheal intubation during hospitalization

ELIGIBILITY:
Inclusion Criteria: Positive SARS-CoV-2 PCR and at least one D-dimer result

Non inclusion Criteria: Below 18 yo

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted at Nancy University Hospital for SARS-CoV-2 infection and with at least one D-dimer result from February 24, 2020 to May 12, 2020.
Sampling Method: Non-Probability Sample
Enrollment: 280 (Actual)
Dates: Start 2020-03-02 (Actual); Primary Completion 2020-08-11 (Actual); Study Completion 2020-08-11 (Actual)

PRIMARY OUTCOMES:
D-dimer trends | From date of admission until the date of first documented thrombosis or date of death from any cause, or date of intubation whichever came first, assessed up to 1 month
  Modifications of D-dimers overtime during the hospitalization

SECONDARY OUTCOMES:
Thrombosis | From date of admission until the date of first documented thrombosis or date of death from any cause, or date of intubation whichever came first, assessed up to 1 month
  Arterial or venous thrombosis
All-cause mortality | From date of admission until the date of first documented thrombosis or date of death from any cause, or date of intubation whichever came first, assessed up to 1 month
  All-cause mortality
Orotracheal intubation | From date of admission until the date of first documented thrombosis or date of death from any cause, or date of intubation whichever came first, assessed up to 1 month
  Orotracheal intubation

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU Nancy, Nancy, France

IPD SHARING:
Plan to Share IPD: No